CLINICAL TRIAL: NCT00620516
Title: Regulatory Requisite Post Marketing Surveillance to Assess the Safety and Efficacy of Spiriva® HandiHaler® (Tiotropium Bromide Inhalation Powder 18mcg, q.d.) in Korean COPD Patients: A 30-Day, Open Label, Non-interventional Study
Brief Title: Tiotropium 18ug Inhalation Capsule Using a Handihaler® Among Korean COPD Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 205.337
Record Dates: First submitted 2008-02-04; First posted 2008-02-21 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a descriptive observational open non-comparative study of the safety and efficacy of tiotropium inhalation capsule given at 18mcg once a day for 30 days among Korean patients with COPD. At Visit 1, patients who are diagnosed as COPD will be prescribed tiotropium inhalation capsule at 18mcg once daily (at the same time). Patients' FEV1 will be assessed before start of treatment (Visit 1) and at the end of the 30 day treatment period (Visit 2). Occurrence of adverse events will also be asked from the patient at the end of the 30 day treatment period. Patients will be informed by the attending physicians to immediately report the occurrence of serious adverse events.

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion Criteria:

Older than 40 years old Diagnosed as COPD No Previous Spiriva administration No Contraindication for Spiriva according to the product label

Exclusion Criteria:

patients with history of hypersensitivity to atropine and its derivatives (e.g. ipratropium oxitropium or any component of this product).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3227
Sampling Method: Probability Sample
Enrollment: 3008 (Actual)
Dates: Start 2004-03; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for this postmarking study is the occurrence of adverse events, anytime during the 30 day study period, which might or might not be connected with the use of Spiriva® 18 mcg inhalation capsule | 30 days

SECONDARY OUTCOMES:
Secondary endpoints include change in post bronchodilator FEV1 and assessment of any change in overall severity of the disease from baseline to the end of 30 day treatment. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (71):
- South Korea (71):
  - Boehringer Ingelheim Investigational Site 1, Busan
  - Boehringer Ingelheim Investigational Site 2, Busan
  - Boehringer Ingelheim Investigational Site 3, Busan
  - Boehringer Ingelheim Investigational Site 4, Busan
  - Boehringer Ingelheim Investigational Site 5, Chugnam
  - Boehringer Ingelheim Investigational Site 6, Chugnam
  - Boehringer Ingelheim Investigational Site 7, Chugnam
  - Boehringer Ingelheim Investigational Site 10, Daegu
  - Boehringer Ingelheim Investigational Site 11, Daegu
  - Boehringer Ingelheim Investigational Site 12, Daegu
  - Boehringer Ingelheim Investigational Site 13, Daegu
  - Boehringer Ingelheim Investigational Site 8, Daegu
  - Boehringer Ingelheim Investigational Site 9, Daegu
  - Boehringer Ingelheim Investigational Site 14, Daejeon
  - Boehringer Ingelheim Investigational Site 15, Daejeon
  - Boehringer Ingelheim Investigational Site 16, Daejeon
  - Boehringer Ingelheim Investigational Site 17, Daejeon
  - Boehringer Ingelheim Investigational Site 18, Daejeon
  - Boehringer Ingelheim Investigational Site 19, Daejeon
  - Boehringer Ingelheim Investigational Site 20, Gangwondo
  - Boehringer Ingelheim Investigational Site 21, Gangwondo
  - Boehringer Ingelheim Investigational Site 22, Gangwondo
  - Boehringer Ingelheim Investigational Site 23, Gangwondo
  - Boehringer Ingelheim Investigational Site 24, Gyeonggido
  - Boehringer Ingelheim Investigational Site 25, Gyeonggido
  - Boehringer Ingelheim Investigational Site 26, Gyeonggido
  - Boehringer Ingelheim Investigational Site 27, Gyeonggido
  - Boehringer Ingelheim Investigational Site 28, Gyeonggido
  - Boehringer Ingelheim Investigational Site 29, Gyeonggido
  - Boehringer Ingelheim Investigational Site 30, Gyeonggido
  - Boehringer Ingelheim Investigational Site 31, Gyeonggido
  - Boehringer Ingelheim Investigational Site 32, Gyeonggido
  - Boehringer Ingelheim Investigational Site 70, Gyeongnam
  - Boehringer Ingelheim Investigational Site 71, Gyeongnam
  - Boehringer Ingelheim Investigational Site 33, Incheon
  - Boehringer Ingelheim Investigational Site 34, Incheon
  - Boehringer Ingelheim Investigational Site 35, Incheon
  - Boehringer Ingelheim Investigational Site 36, Incheon
  - Boehringer Ingelheim Investigational Site 37, Jeonbuk
  - Boehringer Ingelheim Investigational Site 38, Jeonbuk
  - Boehringer Ingelheim Investigational Site 39, Jeonbuk
  - Boehringer Ingelheim Investigational Site 40, Jeonnam
  - Boehringer Ingelheim Investigational Site 41, Jeonnam
  - Boehringer Ingelheim Investigational Site 42, Jeonnam
  - Boehringer Ingelheim Investigational Site 43, Jeonnam
  - Boehringer Ingelheim Investigational Site 44, Jeonnam
  - Boehringer Ingelheim Investigational Site 45, Jeonnam
  - Boehringer Ingelheim Investigational Site 46, Jeonnam
  - Boehringer Ingelheim Investigational Site 69, Jungbuk
  - Boehringer Ingelheim Investigational Site 47, Seoul
  - Boehringer Ingelheim Investigational Site 48, Seoul
  - Boehringer Ingelheim Investigational Site 49, Seoul
  - Boehringer Ingelheim Investigational Site 50, Seoul
  - Boehringer Ingelheim Investigational Site 51, Seoul
  - Boehringer Ingelheim Investigational Site 52, Seoul
  - Boehringer Ingelheim Investigational Site 53, Seoul
  - Boehringer Ingelheim Investigational Site 54, Seoul
  - Boehringer Ingelheim Investigational Site 55, Seoul
  - Boehringer Ingelheim Investigational Site 56, Seoul
  - Boehringer Ingelheim Investigational Site 57, Seoul
  - Boehringer Ingelheim Investigational Site 58, Seoul
  - Boehringer Ingelheim Investigational Site 59, Seoul
  - Boehringer Ingelheim Investigational Site 60, Seoul
  - Boehringer Ingelheim Investigational Site 61, Seoul
  - Boehringer Ingelheim Investigational Site 62, Seoul
  - Boehringer Ingelheim Investigational Site 63, Seoul
  - Boehringer Ingelheim Investigational Site 64, Seoul
  - Boehringer Ingelheim Investigational Site 65, Seoul
  - Boehringer Ingelheim Investigational Site 66, Seoul
  - Boehringer Ingelheim Investigational Site 67, Seoul
  - Boehringer Ingelheim Investigational Site 68, Ulsan